CLINICAL TRIAL: NCT05825651
Title: A Prospective Cohort Study for Long COVID and Health Outcomes in Older Adults in Yunnan, China
Brief Title: Long COVID and Its Associations With Health Outcomes in Older Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Liu Jue, Prof., Peking University
Other Study IDs: NNSF72211540398
Record Dates: First submitted 2023-03-26; First posted 2023-04-24 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Long COVID; COVID-19 Pandemic; Elderly Infection; Vaccine Reaction; Lifestyle Factors; Reinfection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Group with history of COVID-19 infections and vaccines, as well as health-related, behavioral, socioeconomic exposures.
  Interventions: Other: no interventions
- Non-exposure group: Group without history of COVID-19 infections and vaccines, as well as health-related, behavioral, socioeconomic exposures.

INTERVENTIONS:
Other: no interventions — This is an observational study without any intervention.
  Groups: Exposure group

SUMMARY:
The Peking University Health Cohort in Anning, Yunnan (PKUHC-AN) is a prospective cohort study carried out in Anning, Yunnan. The primary aim of this study is to investigate the impact of COVID-19 on older adults' health, and to provide high-quality evidence of real world research for the optimization of prevention and control strategies of COVID-19 and other emerging infectious diseases. Data will be collected regarding health status, history of COVID-19 infections and vaccines, lifestyle and socioeconomic characteristics, as well as the short- and long-term health outcomes.

DETAILED DESCRIPTION:
COVID-19 pandemic attributed to a great number of mortalities around the world in the last 3 years. About 46% of the global population are estimated to have been infected by the omicron variant and its sublineages. Health outcomes post COVID-19 has been of great concern globally since more and more people infected by SARS-CoV-2. Integrated efforts should be made to estimate the incidence of reinfections and long COVID in China, especially among older adults who are vunlerable and susceptible to COVID-19. In view of this, the Peking University Health Cohort Study in Anning, Yunnan aims to investigate the impact of COVID-19 on older adults' health, and to provide high-quality evidence of real world research for the optimization of prevention and control strategies of COVID-19 and other emerging infectious diseases. Data will be collected regarding health status, history of COVID-19 infections and vaccines, lifestyle and socioeconomic characteristics, as well as the short- and long-term health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥60 years
* 2. Resided in Anning in the past half year and have no plan to move out in next 1 year
* 3. Older adults who are willing to participate in this study with informed consent

Exclusion Criteria:

* 1. Unable to answer questions or communicate
* 2. Older adults who are not willing to participate in this study or without informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults aged at least 60 years old living in Anning, Yunnan, China
Sampling Method: Non-Probability Sample
Enrollment: 11527 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of long COVID | From baseline until the date of long COVID symptoms or date of death from any cause, whichever came first, assessed up to 12 months.
  The proportion of participants incurred any symptoms or diagnosed diseases of post-COVID in all infected participants.

SECONDARY OUTCOMES:
Reinfection incidence of COVID-19 | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  The proportion of participants infected by COVID-19 at least 2 times. Measured by trained health professionals.
Cognitive impairment | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  Measured by health professionals using MMSE (Mini-Mental State Exam). The MMSE cognitive screening test is a 30-point questionnaire for analyzing several cognitive functions including memory, orientation, attention, calculation, and language. MMSE is measured on a scale between 0 and 30, where scores of 0-9, 10-20, 21-26, and 27-30 indicate severe, moderate, mild, and normal cognitive function, respectively.
Depression | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  Measured by health professionals using PHQ-9 (Patient Health Questionnaire-9). PHQ-9 provides a score ranging from 0 to 27, where scores of <4, 5-9, 10-14, 15-19, and 20-27 represented no, mild, moderate, moderately severe, and severe depression, respectively.
Medical expenditure | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  Measured by health professionals using self-designed questionnaire about their past month outpatient expenditure and past year inpatient expenditure.
Incidence of catastrophic health expenditure | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  Measured by health professionals using self-designed questionnaire about their households' past year consumption expenditure (including food expenditure, cloths expenditure, transportation expenditure and so on), and calculated as the proportion of households whose out-of-pocket medical expenditure exceed 40% of household non-food expenditure.
Sleep quality | At 3 months, 6 months, 9 months, 1 year after baseline investigation.
  Measured by health professionals using PSQI (Pittsburgh Sleep Quality Index). PSQI reflects sleep for a month, includes 18 items (7 subscales): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction. The range of PSQI global score is 0-21, and a score of >5 or 7 is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Liu, Ph.D, Principal Investigator — Peking University
Locations (1):
- Anning medical community, Kunming, Yunan, China

IPD SHARING:
Plan to Share IPD: No